CLINICAL TRIAL: NCT04041206
Title: A Study on the Microcirculatory Characteristics of Meridian Phenomenon for the Heart and Lung Meridians Based on Patients With Stable Angina Pectoris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Other Study IDs: 2019ZY001-MERIDIAN
Record Dates: First submitted 2019-07-26; First posted 2019-08-01 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Chronic Stable Angina Pectoris
Keywords: meridians; acupuncture; chronic stable angina pectoris; meridian phenomenon; laser doppler
MeSH Terms: interventions — Laser-Doppler Flowmetry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSAP group: This group will include 40 patients with chronic stable angina pectoris (CSAP).
  Interventions: Device: Laser doppler
- Healthy group: This group will include 40 healthy volunteers.
  Interventions: Device: Laser doppler

INTERVENTIONS:
Device: Laser doppler — Laser doppler will be adopted to assess the microcirculatory characteristics of meridian phenomenon for participants in the two groups.
  1. Experimental device: Four-channel laser doppler flowmetry (PeriFlux System 5000, Sweden).
  2. Experimental process: The participants will be allowed to stabilize for 15 minutes in a supine position in the experimental room before formal examination. They are asked to keep silent and normal breath and avoid limb movement during the whole measuring period. The probes will be left at 4 measuring sites. Blood flow curve will be recorded constantly using Perisoft software (PeriFlux, Sweden). Microcirculatory flux in the measuring sites will be calculated [Perfusion units (PU) =concentration of moving blood cells (CMBC)×velocity (V)]. The acupoint microcirculation will be recorded for 5 minutes.
  3. Measurement sites: Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan(LU9) and Chize (LU5) of the Lung meridian

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the microcirculatory characteristics of meridian phenomenon for the Heart and Lung meridians by using laser doppler. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
This study will include 40 patients diagnosed with chronic stable angina pectoris (CSAP) and 40 healthy volunteers. Laser doppler examination will be adopted to assess the microcirculatory characteristics of meridian phenomenon for Heart and Lung meridians in the physiology/pathological state. In addition, by comparing microcirculation in the acupoints along the Heart and Lung meridians, the relative specificity of the two meridians will also be investigated. Primary outcomes will be blood flow curve and blood perfusion units(PU). Furthermore, this study will build standardized techniques and schemes for detecting the microcirculatory characteristics of meridian phenomenon for Heart and Lung. The results of this study could also provide scientific foundation for traditional meridian theories.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for CSAP

1. Patients should meet the diagnostic criteria of coronary heart disease, which includes the following items: 1)confirmed old myocardial infarction (MI), or a history of percutaneous coronary intervention(PCI), or coronary artery bypass grafting; 2)50% or more luminal stenosis in at least one coronary artery or major branch segment confirmed by coronary angiogram or CT angiography; 3) myocardial ischemia indicted by exercise stress radionuclide myocardial imaging; 4) treadmill exercise testing is positive (for male patients);
2. Patients should meet the diagnostic criteria of CSAP and the Canadian Cardiovascular Society(CCS) classification for CSAP is level II or III;
3. The medical history of angina pectoris ≥3 months, with at least 2 episodes per week in the last month;
4. 35 ≤ age ≤65 years, male or female;
5. Patients have clear consciousness and could communicate with others normally;
6. Patients could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent (in the past 3 month) medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. 35 ≤ age ≤65 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for CSAP

1. Patients with acute coronary syndrome (including acute myocardial infarction and unstable angina) and severe arrhythmias (such as severe atrioventricular block, ventricular tachycardia, supraventricular tachycardia, frequent premature beats and premature ventricular contraction);
2. Patients' chest pain is caused by valvular heart disease, hypertrophic cardiomyopathy and dilated cardiomyopathy;
3. Patients' chest pain is caused by non-cardiac disease (such as severe neurosis, climacteric syndrome, cervical spondylosis, and esophageal/pulmonary/chest wall lesions);
4. Patients have concomitant conditions of lung diseases, such as chronic obstructive pulmonary disease (COPD) ;
5. Patients have serious concomitant conditions and and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological and nervous system;
6. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
7. Pregnant or lactating patients;
8. Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have sudden severe diseases during the trial, such as cardiovascular diseases, liver diseases, kidney diseases, urinary diseases and hematological diseases.
2. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
3. Pregnant or lactating participants ;
4. Participants are participating in other trials.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 patients with chronic stable angina pectoris (CSAP) and 40 healthy volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Blood flow curve | 5 minutes
  The blood flow curve could reflect the microcirculatory flux in the measuring sites
Blood perfusion units | 5 minutes
  Perfusion units (PU)=concentration of moving blood cells (CMBC)×velocity (V)

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Ph.D, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hsiu H, Huang SM, Chao PT, Jan MY, Hsu TL, Wang WK, Wang YY. Microcirculatory characteristics of acupuncture points obtained by laser Doppler flowmetry. Physiol Meas. 2007 Oct;28(10):N77-86. doi: 10.1088/0967-3334/28/10/N01. Epub 2007 Sep 18. PMID 17906382
- [Background] Hsiu H, Hsu WC, Chen BH, Hsu CL. Differences in the microcirculatory effects of local skin surface contact pressure stimulation between acupoints and nonacupoints: possible relevance to acupressure. Physiol Meas. 2010 Jun;31(6):829-41. doi: 10.1088/0967-3334/31/6/007. Epub 2010 May 18. PMID 20479520
- [Background] Hsiu H, Hsu WC, Hsu CL, Huang SM, Jan MY, Wang WK, Wang YY. Spectral analysis on the microcirculatory laser Doppler signal at the acupuncture point. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:1084-6. doi: 10.1109/IEMBS.2008.4649348. PMID 19162851
- [Background] Hsiu H, Hsu WC, Hsu CL, Huang SM, Lin YY. Microcirculatory changes by laser Doppler after infrared heating over acupuncture points--relevance to moxibustion. Photomed Laser Surg. 2009 Dec;27(6):855-61. doi: 10.1089/pho.2008.2390. PMID 19698003
- [Background] Hsiu H, Huang SM, Chao PT, Hsu WC, Hsu CL, Jan MY, Wang WK, Wang YY. Study on the microcirculatory blood velocity of acupoint monitored by laser Doppler signal. Annu Int Conf IEEE Eng Med Biol Soc. 2007;2007:959-62. doi: 10.1109/IEMBS.2007.4352451. PMID 18002117
- [Background] Bernard F, Vinet A, Verdant C. Skin microcirculation and vasopressin infusion: a laser Doppler study. Crit Care. 2006;10(2):135. doi: 10.1186/cc4884. PMID 16594988
- [Background] Litscher G, Wang L, Huber E, Nilsson G. Changed skin blood perfusion in the fingertip following acupuncture needle introduction as evaluated by laser Doppler perfusion imaging. Lasers Med Sci. 2002;17(1):19-25. doi: 10.1007/s10103-002-8262-9. PMID 11845364
- [Background] Hsiu H, Hsu WC, Huang SM, Hsu CL, Lin Wang YY. Spectral analysis of the microcirculatory laser Doppler signal at the Hoku acupuncture point. Lasers Med Sci. 2009 May;24(3):353-8. doi: 10.1007/s10103-008-0569-8. Epub 2008 May 27. PMID 18504639
- [Background] Huang T, Wang RH, Zhang WB, Han B, Wang GJ, Tian YY, Zhang YQ. The influence of different methods of acupuncture on skin surface perfusion. J Tradit Chin Med. 2012 Mar;32(1):40-4. doi: 10.1016/s0254-6272(12)60029-6. PMID 22594100

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04041206/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/06/NCT04041206/ICF_001.pdf